CLINICAL TRIAL: NCT00002436
Title: A Randomized Lamivudine (3TC)/Dideoxycytidine (ddC) Double-Blind Multicenter Trial (With Open-Label AZT) to Evaluate the Safety and Efficacy of Low Dose 3TC Administered Concurrently With AZT Versus High Dose 3TC Administered Concurrently With AZT Versus ddC Administered Concurrently With AZT in the Treatment of HIV-1 Infected, AZT-Experienced (>= 24 Weeks) Patients With CD4 Counts of 100-300 Cells/mm3
Brief Title: The Safety and Effectiveness of Three Anti-HIV Drug Combinations in HIV-Infected Patients Who Have Taken AZT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 129C; NUCA 3002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-05

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lamivudine; Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Lamivudine
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To evaluate the safety and efficacy of low and high doses of lamivudine ( 3TC ) in combination with zidovudine ( AZT ) and zalcitabine ( dideoxycytidine; ddC ) in combination with AZT.

PER 02/27/95 AMENDMENT: To evaluate the efficacy and safety of both blinded and open-label combination therapy.

DETAILED DESCRIPTION:
Patients are randomized to one of three treatment arms: low-dose 3TC plus AZT, high-dose 3TC plus AZT, or ddC plus AZT. Treatment continues for 32 weeks, with possible extension to 52 weeks.

PER 02/27/95 AMENDMENT: Patients may continue therapy on AZT and low-dose 3TC on an open-label basis. Open-label therapy continues with follow-up every 8 weeks until intolerable toxicity occurs or study terminates.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity.
* CD4 count 100-300 cells/mm3.
* Prior AZT therapy for 24 or more weeks and currently on AZT.

Exclusion Criteria

Patients with the following prior conditions are excluded:

* History of intolerance to AZT.
* History of grade 2 or worse peripheral neuropathy.

Prior Medication:

Excluded:

* Any prior antiretroviral therapy other than AZT.

Required:

* Concomitant AZT therapy.

Required:

* At least 24 weeks of prior AZT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325

CONTACTS AND LOCATIONS:
Locations (22):
- United States (18):
  - Combat Group, Los Angeles, California
  - San Diego Community Research Group, San Diego, California
  - ViRx Inc, San Francisco, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Louisiana Cardiovascular Research Ctr, New Orleans, Louisiana
  - Boston City Hosp / FGH-1, Boston, Massachusetts
  - Nassau County Med Ctr, East Meadow, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Central Texas Med Foundation, Austin, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Nicholaos Bellos, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Wisconsin Community - Based Research Consortium, Milwaukee, Wisconsin
- Canada (3):
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto Hosp, Toronto, Ontario
  - Montreal Gen Hosp, Montreal, Quebec
- Hosp Regional de Ponce - Area Vieja, Ponce, Puerto Rico